CLINICAL TRIAL: NCT00058695
Title: Evaluation of Single Nucleotide Polymorphism (SNP) in Patients With and Subjects Without Age-Related Macular Degeneration (AMD)
Brief Title: Genetic Factors in Age-Related Macular Degeneration
Status: Terminated | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030155; 03-EI-0155
Record Dates: First submitted 2003-04-11; First posted 2003-04-11 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2015-10-21

CONDITIONS: Macular Degeneration
Keywords: Macualar Degeneration; AMD; Healthy Volunteer; HV
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
This study will examine whether certain polymorphisms (small gene variances) predispose people to develop age-related macular degeneration (AMD). This eye condition affects people over 50 years of age and can cause permanent loss of central vision. The study will examine and compare the frequency of polymorphisms in patients with AMD to that of individuals without AMD. This information will help identify genetic risk factors for the AMD and may lead to the development of more effective treatments.

Patients 50 years of age and older with advanced AMD and healthy normal volunteers may be eligible for this study. All participants will provide an eye health history and will have 10 milliliters (2 teaspoons) of blood drawn from an arm vein. The DNA in the blood will be isolated and tested for certain genes that other research indicates are important in aging and age-related diseases. The normal and polymorphic gene sequences will be identified and compared in patients with AMD and control subjects to determine if any of the polymorphisms are related to development of AMD.

In addition, control subjects will have a routine eye examination, including dilation of the pupils for examination of the back of the eye.

...

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the leading cause of irreversible severe central visual loss older than 50 in the world.1 The incidence and progression of all the features of AMD are known to increase significantly with age.2-4 In a recent study, Klein et al. reported that approximately 15.6% of the US population aged 60 years and older in 2005-2008 had signs of AMD.5 In a study in Iceland, the prevalence of early AMD was 12.4% for those aged 66 to 74 years and 36% for those aged 85 years and older.6 Currently in the United States, advanced AMD affects more than 1.75 million people and the number will increase to 2.95 million by the year 2020.7

Epidemiological studies of genome wide association study (GWAS), candidate gene association, and linkage disequilibrium suggest that AMD has a significant genetic component.7-10 Ample evidence supports the hypothesis that variance of genes involved in DNA repair,11-13 oxidative stress14, 15 and inflammation16-20 play a role in aging and age-related diseases. Many studies have documented the association between polymorphisms in complement factors (CF), oxidative stress, apolipoprotein E (ApoE), mitochondria and chaperone proteins genes and AMD.21-23 Single nucleotide polymorphism (SNP) in ApoE, ApoE or C2/BF may protect AMD. On the other hand, SNP in CFH, AMRS2/HTRA-1 or CX3CR1 gene may increase AMD risk.24 In this study, we would like to test whether the variations of biologically plausible genes (or the modifying genes) listed above are differentially distributed in AMD patients and normal populations. To this end, we choose genes that are believed to play a crucial role in the aging process and will analyze the frequency of SNPs specifically within the coding frames of biologically plausible genes responsible for aging and age-related diseases.

Our aim will be to compare the allelic frequencies of candidate genes listed above in cohorts with AMD to the frequency in normal control subjects without AMD. With this study we hope to identify genetic risk factors that could have functional implications for understanding and treating AMD.

ELIGIBILITY:
* INCLUSION CRITERIA:

AMD Patients (cases):

1. Diagnosis of advanced AMD defined by geographic atrophy and/or choroidal neovascularization with drusen of any size in at least one eye.
2. Age 50 years or older.
3. If sample previously donated in a different study, the patient has given their permission to use their sample (i.e. marked appropriate selection in the informed consent).

Control Patients (controls):

1. Absence of drusen or no more than 5 drusen less than 63 microns, absence of other diagnostic criteria for AMD.
2. Agrees to undergo study examinations.

EXCLUSION CRITERIA:

1. Presence of retinal disease involving the photoreceptors and/or outer retinal layers other than AMD loss such as high myopia, retinal dystrophies, central serous retinopathy, vein occlusion, diabetic retinopathy and uveitis or similar outer retinal diseases that have been present prior to the age of 50.
2. Opacities of the ocular media, limitations of papillary dilation or other problems sufficient to preclude adequate stereo fundus photography. These conditions include occluded pupils due to synechiae, cataracts, vitreous haze and opacities due to ocular diseases.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2003-04-04; Study Completion 2015-10-21

PRIMARY OUTCOMES:
Frequency of SNP | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Nussenblatt, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Tuo J, Ross RJ, Herzlich AA, Shen D, Ding X, Zhou M, Coon SL, Hussein N, Salem N Jr, Chan CC. A high omega-3 fatty acid diet reduces retinal lesions in a murine model of macular degeneration. Am J Pathol. 2009 Aug;175(2):799-807. doi: 10.2353/ajpath.2009.090089. Epub 2009 Jul 16. PMID 19608872
- [Background] Ablikim M, Achasov MN, Albayrak O, Ambrose DJ, An FF, An Q, Bai JZ, Baldini Ferroli R, Ban Y, Becker J, Bennett JV, Bertani M, Bian JM, Boger E, Bondarenko O, Boyko I, Braun S, Briere RA, Bytev V, Cai H, Cai X, Cakir O, Calcaterra A, Cao GF, Cetin SA, Chang JF, Chelkov G, Chen G, Chen HS, Chen JC, Chen ML, Chen SJ, Chen XR, Chen YB, Cheng HP, Chu XK, Chu YP, Cronin-Hennessy D, Dai HL, Dai JP, Dedovich D, Deng ZY, Denig A, Denysenko I, Destefanis M, Ding WM, Ding Y, Dong LY, Dong MY, Du SX, Fang J, Fang SS, Fava L, Feng CQ, Friedel P, Fu CD, Fu JL, Fuks O, Gao Y, Geng C, Goetzen K, Gong WX, Gradl W, Greco M, Gu MH, Gu YT, Guan YH, Guo AQ, Guo LB, Guo T, Guo YP, Han YL, Harris FA, He KL, He M, He ZY, Held T, Heng YK, Hou ZL, Hu C, Hu HM, Hu JF, Hu T, Huang GM, Huang GS, Huang JS, Huang L, Huang XT, Huang Y, Hussain T, Ji CS, Ji Q, Ji QP, Ji XB, Ji XL, Jiang LL, Jiang XS, Jiao JB, Jiao Z, Jin DP, Jin S, Jing FF, Kalantar-Nayestanaki N, Kavatsyuk M, Kloss B, Kopf B, Kornicer M, Kuehn W, Lai W, Lange JS, Lara M, Larin P, Leyhe M, Li CH, Li C, Li C, Li DL, Li DM, Li F, Li G, Li HB, Li JC, Li K, Li L, Li N, Li PR, Li QJ, Li WD, Li WG, Li XL, Li XN, Li XQ, Li XR, Li ZB, Liang H, Liang YF, Liang YT, Liao GR, Lin DX, Liu BJ, Liu CL, Liu CX, Liu FH, Liu F, Liu F, Liu HB, Liu HH, Liu HM, Liu JP, Liu K, Liu KY, Liu PL, Liu Q, Liu SB, Liu X, Liu YB, Liu ZA, Liu Z, Liu Z, Loehner H, Lou XC, Lu GR, Lu HJ, Lu JG, Lu XR, Lu YP, Luo CL, Luo MX, Luo T, Luo XL, Lv M, Ma FC, Ma HL, Ma QM, Ma S, Ma T, Ma XY, Maas FE, Maggiora M, Malik QA, Mao YJ, Mao ZP, Messchendorp JG, Min J, Min TJ, Mitchell RE, Mo XH, Moeini H, Morales Morales C, Moriya K, Muchnoi NY, Muramatsu H, Nefedov Y, Nikolaev IB, Ning Z, Nisar S, Olsen SL, Ouyang Q, Pacetti S, Park JW, Pelizaeus M, Peng HP, Peters K, Ping JL, Ping RG, Poling R, Prencipe E, Qi M, Qian S, Qiao CF, Qin LQ, Qin XS, Qin Y, Qin ZH, Qiu JF, Rashid KH, Redmer CF, Ripka M, Rong G, Ruan XD, Sarantsev A, Schumann S, Shan W, Shao M, Shen CP, Shen XY, Sheng HY, Shepherd MR, Song WM, Song XY, Spataro S, Spruck B, Sun GX, Sun JF, Sun SS, Sun YJ, Sun YZ, Sun ZJ, Sun ZT, Tang CJ, Tang X, Tapan I, Thorndike EH, Toth D, Ullrich M, Uman I, Varner GS, Wang B, Wang D, Wang DY, Wang K, Wang LL, Wang LS, Wang M, Wang P, Wang PL, Wang QJ, Wang SG, Wang XF, Wang XL, Wang YD, Wang YF, Wang YQ, Wang Z, Wang ZG, Wang ZH, Wang ZY, Wei DH, Wei JB, Weidenkaff P, Wen QG, Wen SP, Werner M, Wiedner U, Wu LH, Wu N, Wu SX, Wu W, Wu Z, Xia LG, Xia YX, Xiao ZJ, Xie YG, Xiu QL, Xu GF, Xu QJ, Xu QN, Xu XP, Xu ZR, Xue Z, Yan L, Yan WB, Yan WC, Yan YH, Yang HX, Yang Y, Yang YX, Yang YZ, Ye H, Ye M, Ye MH, Yu BX, Yu CX, Yu HW, Yu JS, Yu SP, Yuan CZ, Yuan WL, Yuan Y, Zafar AA, Zallo A, Zang SL, Zeng Y, Zhang BX, Zhang BY, Zhang C, Zhang CB, Zhang CC, Zhang DH, Zhang HH, Zhang HY, Zhang JQ, Zhang JW, Zhang JY, Zhang JZ, Zhang L, Zhang SH, Zhang XJ, Zhang XY, Zhang Y, Zhang YH, Zhang ZP, Zhang ZY, Zhang Z, Zhao G, Zhao JW, Zhao L, Zhao L, Zhao MG, Zhao Q, Zhao SJ, Zhao TC, Zhao XH, Zhao YB, Zhao ZG, Zhemchugov A, Zheng B, Zheng JP, Zheng YH, Zhong B, Zhou L, Zhou X, Zhou XK, Zhou XR, Zhu K, Zhu KJ, Zhu XL, Zhu YC, Zhu YS, Zhu ZA, Zhuang J, Zou BS, Zou JH; BESIII Collaboration. Observation of a charged charmoniumlike structure Zc(4020) and search for the Zc(3900) in e+e--->pi+pi-hc. Phys Rev Lett. 2013 Dec 13;111(24):242001. doi: 10.1103/PhysRevLett.111.242001. Epub 2013 Dec 10. PMID 24483645
- [Background] Fritsche LG, Chen W, Schu M, Yaspan BL, Yu Y, Thorleifsson G, Zack DJ, Arakawa S, Cipriani V, Ripke S, Igo RP Jr, Buitendijk GH, Sim X, Weeks DE, Guymer RH, Merriam JE, Francis PJ, Hannum G, Agarwal A, Armbrecht AM, Audo I, Aung T, Barile GR, Benchaboune M, Bird AC, Bishop PN, Branham KE, Brooks M, Brucker AJ, Cade WH, Cain MS, Campochiaro PA, Chan CC, Cheng CY, Chew EY, Chin KA, Chowers I, Clayton DG, Cojocaru R, Conley YP, Cornes BK, Daly MJ, Dhillon B, Edwards AO, Evangelou E, Fagerness J, Ferreyra HA, Friedman JS, Geirsdottir A, George RJ, Gieger C, Gupta N, Hagstrom SA, Harding SP, Haritoglou C, Heckenlively JR, Holz FG, Hughes G, Ioannidis JP, Ishibashi T, Joseph P, Jun G, Kamatani Y, Katsanis N, N Keilhauer C, Khan JC, Kim IK, Kiyohara Y, Klein BE, Klein R, Kovach JL, Kozak I, Lee CJ, Lee KE, Lichtner P, Lotery AJ, Meitinger T, Mitchell P, Mohand-Said S, Moore AT, Morgan DJ, Morrison MA, Myers CE, Naj AC, Nakamura Y, Okada Y, Orlin A, Ortube MC, Othman MI, Pappas C, Park KH, Pauer GJ, Peachey NS, Poch O, Priya RR, Reynolds R, Richardson AJ, Ripp R, Rudolph G, Ryu E, Sahel JA, Schaumberg DA, Scholl HP, Schwartz SG, Scott WK, Shahid H, Sigurdsson H, Silvestri G, Sivakumaran TA, Smith RT, Sobrin L, Souied EH, Stambolian DE, Stefansson H, Sturgill-Short GM, Takahashi A, Tosakulwong N, Truitt BJ, Tsironi EE, Uitterlinden AG, van Duijn CM, Vijaya L, Vingerling JR, Vithana EN, Webster AR, Wichmann HE, Winkler TW, Wong TY, Wright AF, Zelenika D, Zhang M, Zhao L, Zhang K, Klein ML, Hageman GS, Lathrop GM, Stefansson K, Allikmets R, Baird PN, Gorin MB, Wang JJ, Klaver CC, Seddon JM, Pericak-Vance MA, Iyengar SK, Yates JR, Swaroop A, Weber BH, Kubo M, Deangelis MM, Leveillard T, Thorsteinsdottir U, Haines JL, Farrer LA, Heid IM, Abecasis GR; AMD Gene Consortium. Seven new loci associated with age-related macular degeneration. Nat Genet. 2013 Apr;45(4):433-9, 439e1-2. doi: 10.1038/ng.2578. Epub 2013 Mar 3. PMID 23455636